CLINICAL TRIAL: NCT07328945
Title: Patient-derived Tumor-like Cell Cluster Model-based Precision Treatment Strategy on Non-small Cell Lung Cancer: a Prospective, Observational Study
Brief Title: Patient-derived Tumor-like Cell Cluster Model-based Precision Treatment Strategy on Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Deputy Director of MD. PhD. Program in Thoracic Surgery, Secretary of the party committee of Shanghai Pulmonary Hospital, Tongji University School of Medicine, Shanghai, China, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: STAR015
Record Dates: First submitted 2024-06-03; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Patient-derived Tumor-like Cell Cluster; Precision Treatment Strategy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Malignant pleural effusion or tumour puncture sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTC drug-testing high response group
  Interventions: Diagnostic Test: PTC predicts the response to drug therapy in lung cancer patients
- PTC drug-testing low response group
  Interventions: Diagnostic Test: PTC predicts the response to drug therapy in lung cancer patients

INTERVENTIONS:
Diagnostic Test: PTC predicts the response to drug therapy in lung cancer patients — a Prospective, Observational Study

SUMMARY:
This trial is a prospective, observational study of non-small cell lung cancer that aims to evaluate the feasibility, preliminary efficacy and safety of patient-derived tumor-like cell cluster model in guiding the precision treatment strategy.

DETAILED DESCRIPTION:
The investigators have established a precision treatment strategy, that select immunotherapy drugs or chemotherapeutic drugs or targeted drugs based on information from PTCs drug-screening or/and bioinformatic prediction. In this study, the investigators are going to exploit this strategy for the precision treatment of advanced stage non-small cell lung cancer (NSCLC). The investigators will evaluate the feasibility, safety and preliminary efficacy via collecting the indexes comprising clinical presentation, results of imaging examination, objective response rate, progression free survival etc. In addition, investigators will investigate the changes in the tumor immune microenvironment during drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years and ≤80 years;
2. Non-small cell lung cancer diagnosed by pathology (including histology or cytology);
3. Having measurable lesions (according to RECIST 1.1 criteria, the long diameter of CT scan of tumour lesion is ≥10mm, the short diameter of CT scan of lymph node lesion is ≥15mm, the thickness of scanning layer is not more than 5mm, and the measurable lesion has not received local treatment such as radiotherapy, cryotherapy, etc.);
4. ECOG PS: 0-2 points;
5. Expected survival ≥ 3 months;
6. Adequate hepatic function, defined as total bilirubin levels ≤ 1.5 times the upper limit of normal (ULN) and alanine aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times the ULN in all patients;
7. Adequate renal function, defined as creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula);
8. Adequate coagulation function, defined as International Normalised Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN; if the subject is on anticoagulant therapy, as long as the INR/PT is within the range formulated for the anticoagulant drug;
9. For female subjects of childbearing potential, a negative urine or serum pregnancy test should be presented within 3 days prior to receiving the first dose of study drug, or a blood pregnancy test will be requested if the urine pregnancy test result cannot be confirmed as negative;
10. If there is a risk of conception, male and female patients are required to use highly effective contraception (i.e., a method with a failure rate of less than 1% per year) for at least 180 days after discontinuation of trial treatment; NOTE: Abstinence is acceptable as a method of contraception if abstinence is the subject's usual lifestyle and preferred method of contraception;
11. Subjects voluntarily enroll in the study, sign a written informed consent prior to the implementation of any trial-related process, are compliant, and cooperate with follow-up visits.

Exclusion Criteria:

1. Currently participating in an interventional clinical study treatment, or have received another investigational drug or investigational device within 4 weeks prior to the first dose;
2. Have received a proprietary medicine with an anti-tumor indication or an immunomodulatory drug (thymidine, interferon, interleukin, etc.) within 2 weeks prior to the first dose, or have received major surgical treatment within 3 weeks prior to the first dose;
3. Presence of active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction and peritoneal metastases requiring clinical intervention;
4. Known or screening test findings of active central nervous system (CNS) metastases and/or carcinomatous meningitis;
5. Has received a solid organ or blood system transplant;
6. Class III-IV congestive heart failure (New York Heart Association classification) with poorly controlled and clinically significant arrhythmias;
7. Any arterial thrombosis, embolism or ischemia such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack within 6 months prior to enrolment for treatment. History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism within 3 months prior to enrolment (implantable IV port or catheter-derived thrombosis, or superficial venous thrombosis are not considered "serious" thromboembolism);
8. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency) are not considered systemic therapy;
9. Patients requiring long-term systemic corticosteroids. Patients requiring intermittent use of bronchodilators, inhaled corticosteroids, or locally injected corticosteroids due to COPD, asthma may be enrolled;
10. Diagnosis of other malignancy within 5 years prior to the first dose, excluding radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ, and if diagnosed with other malignancy or lung cancer more than 5 years prior to the dose, pathological or cytological diagnosis of recurrent metastatic lesions is required;
11. Known psychiatric or substance abuse conditions that may have an impact on compliance with the trial requirements;
12. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive), known syphilis infection (syphilis antibody positive), active tuberculosis;
13. untreated active hepatitis B; Note: Subjects with hepatitis B who meet the following criteria are also eligible for enrolment: HBV viral load must be <1000 copies/ml (200 IU/ml) or below the lower limit of detection prior to the first dose of drug, and subjects should be treated with anti-HBV therapy to avoid viral reactivation for the entire duration of the study chemotherapeutic agent treatment. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required but close monitoring of viral reactivation is needed;
14. Subjects with active HCV infection (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
15. Live vaccination within 30 days prior to the first dose; NOTE: It is permissible to receive injectable inactivated viral vaccine against seasonal influenza; however, it is not permissible to receive live attenuated influenza vaccine administered intranasally;
16. The presence of abnormal results from a medical history, disease, treatment, or laboratory that could interfere with the results of the trial, prevent the subject from participating in the study throughout its duration, or where participation in the study is not, in the opinion of the Investigator, in the best interest of the subject;
17. Local or systemic disease, or secondary reactions to cancer, not due to malignancy and which may result in a higher medical risk and/or uncertainty in the evaluation of survival.
18. Persons who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer diagnosed by pathology (including histology or cytology)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Concordance Rate between PTC drug-sensitivity results and clinical response | 6 months
  Clinical response is evaluated according to RECIST 1.1 criteria. Concordance rate is defined as the percentage of participants whose clinical response (Complete Response or Partial Response) matches the predicted sensitivity by the PTC assay.

SECONDARY OUTCOMES:
Progression free survival | 3 years
  The progression free survival between PTC drug-testing high group with PTC drug-testing low group
Difference in Proportion of Tumor-Infiltrating Immune Cell Subsets (e.g., T cells, B cells, Macrophages). | 6 months
  Evaluated by single-cell RNA sequencing (scRNA-seq) or transcriptomic analysis on samples (pleural effusion, biopsy, etc.). Data will be reported as the percentage of specific immune cell types (e.g., CD4+, CD8+ T cells, Tregs, M1/M2 macrophages) relative to total cells, comparing the PTC drug-testing high group with the low group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided